CLINICAL TRIAL: NCT01853241
Title: Prospective Randomized Trial of Anterograde Single Balloon Versus Spirus Enteroscopy in Patients With Suspected Small Bowel Disease
Brief Title: Prospective Randomized Trial of Anterograde Single Balloon Versus Spirus Enteroscopy
Status: Terminated | Type: Observational
Why Stopped: SE system by Spirus Medical withdrawn from market in 2011
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Patrick Okolo, MD, Chief, Gastrointestinal Endoscopy; Associate Professor of Medicine, Johns Hopkins University
Other Study IDs: NA_00031000JHU; NA_00031000 (Other: Johns Hopkins Medicine)
Record Dates: First submitted 2013-05-10; First posted 2013-05-14 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-05

CONDITIONS: Gastrointestinal Hemorrhage; Inflammatory Bowel Disease; Gastrointestinal Neoplasms
Keywords: small intestine; endoscopy, gastrointestinal
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Inflammatory Bowel Diseases; Gastrointestinal Neoplasms | interventions — Single-Balloon Enteroscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Single balloon: Single Balloon Enteroscopy
  Interventions: Procedure: Single Balloon
- Spirus: Spirus Enteroscopy
  Interventions: Procedure: Spirus

INTERVENTIONS:
Procedure: Single Balloon — All patients in this group will undergo single balloon enteroscopy
  Other Names: Single Balloon Enteroscopy
  Groups: Single balloon
Procedure: Spirus — All patients in this group will undergo Spirus Enteroscopy
  Other Names: Spirus Enteroscopy
  Groups: Spirus

SUMMARY:
The small bowel is poorly suited to standard endoscopy techniques due to its anatomical differences from the colon and the upper gastrointestinal tract. The small bowel has an average length of 6.7 m, with a free mesentery that resists standard "push to advance" endoscopy techniques. New developments in overtubes, which are placed over an enteroscope, have revolutionized doctors ability to deeply intubate the small bowel. Three types of 'augmented' enteroscopy, double balloon enteroscopy (DBE), single balloon enteroscopy (SBE) and spiral enteroscopy (SE), have been developed. Although studies have been performed on these individual techniques, there are no studies comparing SBE and SE, the two techniques used in Johns Hopkins.

The investigators propose performing a prospective, randomised trial, to assess the differences between these two techniques. The question of what differences there are between these two techniques, in terms of depth of insertion, diagnostic and therapeutic yields, time required for the procedure and the sedation requirements, are important questions to answer, and depending on the results, would affect the investigators approach to patients with small bowel disease.

DETAILED DESCRIPTION:
We currently perform both spiral enteroscopy (SE) and single balloon enteroscopy (SBE) in Johns Hopkins Hospital. The decision as to which procedure to use is determined by the endoscopist performing the procedure, with currently approximately 60% being performed with SE and 40% performed with SBE. We wish to perform a prospective, randomised trial, to assess the differences between these two procedures. The question of what differences there are between these two techniques, in terms of depth of insertion, diagnostic and therapeutic yields, time required for the procedure and the sedation requirements, are important questions to answer, and depending on the results, would affect the investigators approach to patients with small bowel disease.

The small bowel is poorly suited to standard endoscopy techniques due to its anatomical differences from the colon and the upper gastrointestinal tract. The small bowel has an average length of 6.7 m, with a free mesentery that resists standard "push to advance" endoscopy techniques. New developments in overtubes, which are placed over an enteroscope, have revolutionized the investigators ability to deeply intubate the small bowel. The first of these new techniques to be described was double balloon enteroscopy (DBE) (Fujinon, Wayne, NJ) in 2001. The next development was single balloon enteroscopy (SBE) (Olympus America, Center Valley PA), an iteration of DBE that simply forgoes the second balloon at the tip of the endoscope, and also allows for deep enteroscopy which has been available in the United States since 2007. Spiral enteroscopy (SE) was introduced soon after SBE in 2007, and consists of a spiral overtube (Spirus Medical Inc., Stoughton, Massachusetts, USA) which pleats the small bowel onto the enteroscope.

DBE has the largest amount of published data, with more than 1370 patients and 2591 examinations. Data regarding the efficacy of SBE and SE are more limited than DBE. SBE and SE have only been available in the United States since 2007, and therefore have less published data than DBE. There are two published series of SBE, with several more publications in abstract form. A total of 362 cases have been reported, with diagnostic yields ranging between 30% to 76%, with therapeutic intervention performed in up to 55%. There are 6 reports of SE procedures, with one large series of 1750 cases documenting side effects of SE. The overall diagnostic yield ranged from 24% to 51% with similar treatment success rates. SBE has been compared with DBE in patients with suspected small bowel disease in three studies reported in abstract form. SE has been compared with push enteroscopy and DBE, however there have been no studies comparing SBE and SE.

The risks associated with augmented enteroscopy (DBE, SBE, SE) are similar to those associated with routine endoscopy and include sedation-related complications, aspiration pneumonia, and respiratory infections. In addition, there have been complications specifically related to augmented enteroscopy. Abdominal discomfort can occur due to trapped gas. DBE has been associated with intestinal cramping in 2% to 20% of patients. The use of CO2, which the investigators routinely use in Johns Hopkins, decreases post procedure abdominal cramping. Minor small bowel contusion can occur. The incidence of gastrointestinal haemorrhage does not seem to be increased in augmented enteroscopy compared with standard endoscopic procedures. Pancreatitis occurred in 6 (0.2%) of cases reported in a multicenter United States study of DBE. There have been no reports of pancreatitis associated with SBE or SE enteroscopy. Intestinal perforation is a rare but serious event. Perforation has been reported in 5 (0.2%) of 2591 DBE examinations. In SBE, one perforation was reported in a series of 37 patients, with a case report of a perforation in a patients with jejuna ulceration from metastatic adenocarcinoma of unknown primary. A mucosal tear, requiring endoscopic clip esophageal or gastric perforation, severe bleeding requiring transfusion, cardio-pulmonary arrests or deaths. There were 7 (0.4%) severe complications. Six were small bowel perforations (0.34%).

In Johns Hopkins there has been one perforation using SBE and one using SE one of which occurred in a patient with small bowel Crohns disease (SBE) and the other in a patient with altered anatomy (SE) (personal communication Dr PI Okolo). This latter group of patients are known to be at increased risk of perforation during endoscopic procedures and will be excluded from this study. There have had no other serious complication associated with either SE or SBE enteroscopy. All of the individuals who will participate in this study are already scheduled to have an augmented enteroscopy. Therefore, there is no additional risk incurred by the patient by participating in this study, over and above the risk of an augmented enteroscopy which is part of the routine clinical care for these patients.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old
* Referred to Johns Hopkins Hospital for anterograde augmented enteroscopy to assess for small bowel disease

Exclusion Criteria:

* Patients who are unable to give informed consent
* Women who are pregnant
* Inability to tolerate sedated endoscopy due to cardio-pulmonary instability or other contraindication to endoscopy
* Patients who require retrograde enteroscopy as determined by the principle investigator
* Patients with altered small bowel anatomy (i.e. Roux-en-Y anastomosis, Bilroth II anatomy)
* Cirrhosis
* Esophageal stricture
* Uncorrected coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to our center for anterograde augmented enteroscopy for the assessment of suspected small disease
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2010-05; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Comparison of the depth of insertion into the small bowel of SBE compared with SE from the pylorus. | At the time of procedure
  The depth of insertion was defined as the maximum distance the enteroscope was inserted past the pylorus. In SBE, the endoscopist estimates in 10cm increments from 0 to 40 cm the length of small bowel released during each insertion of the overtube and pulling back of the enteroscope and overtube. The net advancement is defined as the DMI for SBE. For SE the DMI is calculated by counting the length of bowel examined in 10-cm increments upon withdrawal of the enteroscope and overtube.

SECONDARY OUTCOMES:
Comparison of the complication rate between the two techniques. | 7 days of procedure
  Patients were contacted by telephone within 1 week of the procedure. Immediate and short term complications were recorded. Major complications were defined as deep laceration, perforation, significant bleeding requiring blood products, pancreatitis, or hospital admission related to the procedure. Minor complications were defined as mild to moderate mucosal trauma (score 1-3), sore throat less than 72 hours in duration, abdominal discomfort lasting less than 48 hours in duration, or mild nausea or vomiting.
  Mucosal trauma was evaluated upon withdrawal of the enteroscope. Pain was assessed on a 10 point visual analogue scale before and after the procedure. Patients underwent a telephone interview within 7 days of the procedure where the type and severity of side effects and complications were assessed
Comparison of the diagnostic yield between the two techniques. | immediate
  Diagnostic yield was defined as the number of patients who had a diagnosis confirmed with enteroscopy.
Comparison of the therapeutic yield between the two techniques. | immediate
  Therapeutic yield was defined as the number of patients who required a intervention at the time of enteroscopy
A comparison of the mean adjusted diagnostic procedure time | immediate
  This is calculated by for all procedures: total time minus therapy time.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Okolo, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Background] Hartmann D, Eickhoff A, Tamm R, Riemann JF. Balloon-assisted enteroscopy using a single-balloon technique. Endoscopy. 2007 Feb;39 Suppl 1:E276. doi: 10.1055/s-2007-966616. Epub 2007 Oct 24. No abstract available. PMID 17957636
- [Background] Akerman PA, Agrawal D, Cantero D, Pangtay J. Spiral enteroscopy with the new DSB overtube: a novel technique for deep peroral small-bowel intubation. Endoscopy. 2008 Dec;40(12):974-8. doi: 10.1055/s-0028-1103402. Epub 2008 Dec 8. PMID 19065477
- [Background] Tsujikawa T, Saitoh Y, Andoh A, Imaeda H, Hata K, Minematsu H, Senoh K, Hayafuji K, Ogawa A, Nakahara T, Sasaki M, Fujiyama Y. Novel single-balloon enteroscopy for diagnosis and treatment of the small intestine: preliminary experiences. Endoscopy. 2008 Jan;40(1):11-5. doi: 10.1055/s-2007-966976. Epub 2007 Dec 4. PMID 18058613
- [Background] Kawamura T, Yasuda K, Tanaka K, Uno K, Ueda M, Sanada K, Nakajima M. Clinical evaluation of a newly developed single-balloon enteroscope. Gastrointest Endosc. 2008 Dec;68(6):1112-6. doi: 10.1016/j.gie.2008.03.1063. Epub 2008 Jul 2. PMID 18599052
- [Background] Akerman PA, Cantero D. Spiral enteroscopy and push enteroscopy. Gastrointest Endosc Clin N Am. 2009 Jul;19(3):357-69. doi: 10.1016/j.giec.2009.04.001. PMID 19647645
- [Background] Mehdizadeh S, Ross A, Gerson L, Leighton J, Chen A, Schembre D, Chen G, Semrad C, Kamal A, Harrison EM, Binmoeller K, Waxman I, Kozarek R, Lo SK. What is the learning curve associated with double-balloon enteroscopy? Technical details and early experience in 6 U.S. tertiary care centers. Gastrointest Endosc. 2006 Nov;64(5):740-50. doi: 10.1016/j.gie.2006.05.022. PMID 17055868
- [Background] Heine GD, Hadithi M, Groenen MJ, Kuipers EJ, Jacobs MA, Mulder CJ. Double-balloon enteroscopy: indications, diagnostic yield, and complications in a series of 275 patients with suspected small-bowel disease. Endoscopy. 2006 Jan;38(1):42-8. doi: 10.1055/s-2005-921188. PMID 16429354
- [Background] Gerson LB. Outcomes associated with deep enteroscopy. Gastrointest Endosc Clin N Am. 2009 Jul;19(3):481-96. doi: 10.1016/j.giec.2009.04.007. PMID 19647653
- [Background] Vincent JR. [The "Mobile Dental Health Clinic of the South-West" (2)]. J Dent Que. 1991 Jul-Aug;28:341-7. French. PMID 1960245